CLINICAL TRIAL: NCT01341665
Title: Subclassification of the Syndrome of Inappropriate Antidiuresis Via Copeptin - What is the Genesis of ADH-independent SIADH?
Brief Title: Subclassification of the Syndrome of Inappropriate ADH Secretion
Status: Completed | Type: Observational
Sponsor: University of Wuerzburg (Other)
Responsible Party: Prof. Dr. Bruno Allolio, Department of Endocrinology and Diabetes, University of Wuerzburg
Other Study IDs: 5/08
Record Dates: First submitted 2011-04-21; First posted 2011-04-26 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-04

CONDITIONS: Hyponatremia
Keywords: hyponatremia; SIADH; copeptin
MeSH Terms: conditions — Hyponatremia; Inappropriate ADH Syndrome; Diabetes Insipidus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to evaluate the different types of osmotic dysregulation in patients with Syndrome of Inappropriate ADH (SIADH) and, hence, to analyze the pathophysiology of SIADH.

These types will be characterized by measurement of AVP and copeptin while performing an osmotic stimulation with infusion of hypertonic saline.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years,
* hyponatremia < 132 mmol/L
* SIADH

Exclusion Criteria:

* age < 18 years
* cerebral metastases
* serum sodium > 132mmol/L

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with chronic hyponatremia (> 3 days) due to SIADH in university hospital in wuerzburg
  healthy control subjects with normonatremia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Allolio, MD, Study Chair — Ethical commitee
Locations (1):
- University of Wuerzburg, Würzburg, Bavaria, Germany